CLINICAL TRIAL: NCT01903707
Title: Cognitive Remediation in Schizophrenia: Effects on Brain Structure, Brain Function and Social Outcome.
Brief Title: Cognitive Remediation in Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Gary Donohoe, Associate Professor, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRT001
Record Dates: First submitted 2013-07-02; First posted 2013-07-19 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Schizophrenia; Psychosis
Keywords: Schizophrenia; Psychosis; Cognitive deficits
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Remediation Therapy (Experimental): Participants will undertake approximately 30 minutes of computerized CRT training for 8 weeks, 5 days per week. They will meet a therapist once per week to discuss any difficulties, help motivation.
  Interventions: Other: Cognitive Remediation Therapy
- Placebo Comparator (Placebo Comparator): Participants will meet therapist once per week but will not undertake the Computerized Cognitive remediation training.
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Other: Cognitive Remediation Therapy — Computerised training undertaken for approximately 30 minutes per day, 5 days per week for 8 weeks
  Other Names: CRT
  Arms: Cognitive Remediation Therapy
Other: Placebo comparator — Participant meets the therapist once per week but does not carry out the CRT intervention. (Participants are subsequently offered the chance to carry out the CRT intervention post study if they so wish).
  Other Names: No intervention
  Arms: Placebo Comparator

SUMMARY:
The aim of this project is to undertake a randomized placebo controlled trial of cognitive remediation therapy (CRT) that focuses on working memory training in a sample of community based patients with chronic schizophrenia or other psychoses.

Cognitive deficits are a problem for many people with schizophrenia. This study will use computerized cognitive remediation training (which the participant can carry out at home) over a period of a few months.

DETAILED DESCRIPTION:
The aim of this project is to undertake a randomized placebo controlled trial of cognitive remediation therapy (CRT) that focuses on working memory training in a sample of community based patients with schizophrenia. Pre and Post neuropsychological assessment and Magnetic Resonance Imagery (MRI) will be used to determine the effects of CR training on

1. Neuropsychological performance
2. Brain Structure using voxel-based morphometry (VBM)
3. Brain function using functional MRI (fMRI)
4. Social and occupational functioning

The cognitive remediation intervention is a computerised programme whose training level is dynamically varied to suit participants individual ability level. Motivation to learn and generalization to real world function are a particular focus of the intervention and are supported with ongoing therapist interaction in addition to personal training.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia
* History of Psychosis
* Subjective difficulties with memory or concentration
* Aged 18-60 Years

Exclusion Criteria:

* History of head injury resulting in loss of consciousness
* Substance misuse in the last 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline neuropsychological performance | Directly following study treatment period
  A battery of neuropsychological tests will be used at baseline and the same tests used directly after the intervention to measure changes in attention and memory. Tests include Wechsler Adult intelligence scale-III, Wechsler Memory Scale-III, Stroop test, Wisconsin card sorting task and measures of spatial working memory.

SECONDARY OUTCOMES:
Change from baseline neuropsychological performance at 3 to 6 months post intervention | 3 to 6 months post study treatment period
  A battery of neuropsychological tests will be used at baseline and the same tests used at 3 months post intervention to measure changes in attention and memory. Tests include Wechsler Adult intelligence scale-III, Wechsler Memory Scale-III, Stroop test, Wisconsin card sorting task and measures of spatial working memory.
Changes from baseline in brain activation during working memory testing | Directly post study treatment period
  Changes from baseline in brain activation during working memory testing will be measured using fMRI
Change from baseline in grey matter volume | Directly following study treatment period
  Changes in grey matter volume from baseline will be measured at 3 months post intervention using voxel based morphometry.

OTHER OUTCOMES:
Changes in social and occupational functioning | Directly following study treatment period
  Social and occupational function will be measured at baseline and the same tests used directly following intervention. Standardised measures will be used including ILS (Independent Living Scales) and the UCSD performance skills assessment brief version(UPSA-B)
Change from baseline in social and occupational functioning 3 to 6 months post intervention | 3 to 6 months post study treatment period
  Social and occupational function will be measured at baseline and the same tests used directly following intervention. Standardised measures will be used including ILS (Independent Living Scales) and the UCSD performance skills assessment brief version(UPSA-B)

CONTACTS AND LOCATIONS:
Overall Officials: Gary J Donoghoe, DClin Psych PhD, Principal Investigator — Trinity College Dublin, Ireland
Locations (1):
- Department of Psychiatry, Trinity Centre for Health Sciences, St James Hospital, James St., Dublin, Dublin, Ireland